CLINICAL TRIAL: NCT00110474
Title: Efficacy and Safety of Glucosamine Sulfate Versus a Pure Analgesic (Acetaminophen/Paracetamol) and Placebo in Patients Suffering From Osteoarthritis of the Knee
Brief Title: Glucosamine Unum In Die [Once A Day] Efficacy (GUIDE) Trial: Glucosamine Sulfate in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rottapharm (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JN151198
Record Dates: First submitted 2005-05-09; First posted 2005-05-10 (Estimated); Last update posted 2006-09-19 (Estimated); Status verified 2006-09

CONDITIONS: Knee Osteoarthritis
Keywords: Glucosamine sulfate; Osteoarthritis; Acetaminophen; Paracetamol; Clinical trial
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Glucosamine; Acetaminophen

INTERVENTIONS:
Drug: Glucosamine sulfate
Drug: Acetaminophen

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of glucosamine sulfate versus placebo on the symptoms of knee osteoarthritis after 6 months of treatment, using acetaminophen as a reference symptomatic medication.

DETAILED DESCRIPTION:
Osteoarthritis is a common degenerative joint disease, affecting a large proportion of the general population. Its severity is progressive and often requires long-term treatment courses.

Medications for osteoarthritis may affect symptoms (pain and function limitation) and/or modify joint structure.

Pharmacological agents usually employed to treat symptoms generally include unspecific drugs such as pure analgesics and non-steroidal antiinflammatory drugs (NSAIDs), as well as compounds that are possibly disease specific, since they probably interact with some of the osteoarthritis pathogenetic factors: glucosamine sulfate is one of these agents.

Glucosamine sulfate has recently attracted the attention of the scientific community and of patients, because two long-term (3 years) clinical trials in comparison with placebo, showed that this is the first agent able to retard the progression of anatomic joint structure changes in knee osteoarthritis, besides controlling the progression of symptoms.

Earlier studies had shown that glucosamine sulfate is effective in relieving the symptoms of osteoarthritis also over shorter treatment courses (few weeks or months), in comparison with placebo. In addition, glucosamine sulfate efficacy in short studies was at least comparable to that of unspecific symptomatic medications such as conventional NSAIDs, whilst being better tolerated. However, all practice guidelines for the treatment of osteoarthritis suggest acetaminophen (paracetamol) as the oral analgesic to try first and, if successful, the preferred long-term symptomatic medication.

This trial was therefore designed to confirm the efficacy of glucosamine sulfate in comparison with placebo and to assess its relative value compared with acetaminophen. In fact, superiority of a well tolerated drug such as glucosamine sulfate and with the long-term treatment potential shown in other trials, may represent a major therapeutic advantage.

The treatment has a duration of 6 months, that is believed to be the minimum length to assess the effects of a symptomatic medication in osteoarthritis.

The study is performed according to a multicenter, randomised, placebo- and reference-controlled, double-blind (double-dummy), parallel group, prospective design.

The sample size has been calculated on the basis of the expected efficacy of the test drug on the primary outcome (Lequesne index).

Following a screening visit and a short baseline period to check adherence to the inclusion/exclusion criteria, a total of at least 300 patients with knee osteoarthritis are randomised to receive either oral glucosamine sulfate soluble powder 1500 mg once-a-day, or acetaminophen tablets 1000 mg three times a day (total 3g/day, as recommended in Europe), or placebo, for 6 months. The rescue medication for flare episodes consists of the standardized use (according to specific instructions given to the patients) of ibuprofen 400 mg tablets, whose consumption is recorded in a patient daily diary.

The primary efficacy outcome measure is represented by the change in the Lequesne algo-functional index (assessed at clinic visits) after 6 months in the intention-to treat population, analysed by the General Linear Model (GLM) procedure for ANOVA, with Dunnet's pairwise comparisons versus placebo. Efficacy in patients completing treatment according to the protocol (per-protocol completers) will be also assessed. Secondary efficacy outcome measures include the changes in the WOMAC index and the calculation of the proportion of patients that can be defined responders to treatment according to the Osteoarthritis Research Society International (OARSI) criteria (2000). The use of the rescue medication is also assessed.

Safety is assessed by reporting of adverse events and by routine laboratory tests.

The glucosamine sulfate substance used in this trial (crystalline glucosamine sulfate) is a prescription drug in Europe and elsewhere, mostly used in its 1500 mg powder for oral solution formulation to be administered once daily. This is the substance/formulation that was effective and safe in the vast majority of glucosamine clinical trials, including the long-term, 3-year studies.

Differently than in Europe and other countries, glucosamine formulations are marketed in the United States as dietary supplements. They include glucosamine sulfate substances different than the original prescription preparation, other glucosamine salts (mainly glucosamine hydrochloride), and are administered according to different dosage schemes (mainly as oral solid formulations that provide a total 1500 mg dose, but divided in three daily intakes, t.i.d.). In clinical trials conducted so far, these formulations failed to show the same efficacy of the original glucosamine sulfate prescription preparation.

The present study uses therefore the original prescription crystalline glucosamine sulfate given once-a-day (unum-in-die, u.i.d.) and it is therefore named the Glucosamine Unum In Die Efficacy (GUIDE) Trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of knee osteoarthritis according to the clinical and radiological criteria of the American College of Rheumatology (ACR), with minimum symptom severity/characteristics

Exclusion Criteria:

* Standard exclusions apply

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2000-05; Study Completion 2002-12

PRIMARY OUTCOMES:
Lequesne Index

SECONDARY OUTCOMES:
WOMAC Index
OARSI Responder Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Herrero-Beaumont, MD, Study Director — Fundacíón Jiménez Díaz - Madrid - Spain
Locations (13):
- Portugal (3):
  - Hospital Universitario de Coimbra, Coimbra
  - Hospital Egaz Moniz, Lisbon
  - Hospital Conde do Bertiandos, Ponte de Lima
- Spain (10):
  - Complejo Hospitalario Juan Canalejo, A Coruña
  - Hospital Clinic, Barcelona
  - Hospital del Mar, Barcelona
  - Completo Hospitalario de Ciudad Real, Ciudad Real
  - Hospital Donostia, Donostia / San Sebastian
  - Fundacíón Jiménez Díaz, Madrid
  - Hospital de La Pricesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Nuestra Señora de Valme, Seville
  - Hospital Dr. Peset, Valencia

REFERENCES:
- [Result] Herrero-Beaumont G, Román JA, Trabado MC, Blanco FJ, Benito P, Martin-Mola E, et al. Effects of glucosamine sulfate on 6-month control of knee osteoarthritis symptoms vs. placebo and acetaminophen: results from the Glucosamine Unum In Die Efficacy (GUIDE) trial [abstract]. Arthritis Rheum 2005;9 Suppl: 1203.
- [Derived] Herrero-Beaumont G, Ivorra JA, Del Carmen Trabado M, Blanco FJ, Benito P, Martin-Mola E, Paulino J, Marenco JL, Porto A, Laffon A, Araujo D, Figueroa M, Branco J. Glucosamine sulfate in the treatment of knee osteoarthritis symptoms: a randomized, double-blind, placebo-controlled study using acetaminophen as a side comparator. Arthritis Rheum. 2007 Feb;56(2):555-67. doi: 10.1002/art.22371. PMID 17265490